

| To | Tsang Wai Nam (Department of Rehabilitation Sciences) TSANG Wing Hong Hector, Chair, Departmental Research Committee | | |
|---|---|---|---|
| From | | | |
| Email | rshtsang@inet.polyu.edu.hk | Date | 03-Oct-2018 |

## Application for Ethical Review for Teaching/Research Involving Human Subjects

I write to inform you that approval has been given to your application for human subjects ethics review of the following project for a period from 29-Oct-2018 to 30 Sep 2020.

Project Title: The effects of sitting Tai Chi training on balance, eye-hand

coordination, physical fitness and quality of life in non-

ambulatory subjects with Parkinson disease

**Department:** Department of Rehabilitation Sciences

Principal Investigator: Tsang Wai Nam

Please note that you will be held responsible for the ethical approval granted for the project and the ethical conduct of the personnel involved in the project. In the case of the Co-PI, if any, has also obtained ethical approval for the project, the Co-PI will also assume the responsibility in respect of the ethical approval (in relation to the areas of expertise of respective Co-PI in accordance with the stipulations given by the approving authority).

You are responsible for informing the Departmental Research Committee in advance of any changes in the proposal or procedures which may affect the validity of this ethical approval.

You will receive separate email notification should you be required to obtain fresh approval.

TSANG Wing Hong Hector

Chair

Departmental Research Committee